CLINICAL TRIAL: NCT03832374
Title: Study of the Association Between Subtypes of Anti Citrullinated Peptide Antibodies and Lung Damage in Rheumatoid Arthritis in the West Indies
Brief Title: Association Between Subtypes of Anti Citrullinated Peptide Antibodies and Lung Damage in Rheumatoid Arthritis
Acronym: ACPPPA
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 15/E/27
Record Dates: First submitted 2018-10-29; First posted 2019-02-06 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Descriptive

SUMMARY:
Rheumatoid arthritis is a genuine systemic disease associated with diffuse interstitial pneumopathy and bronchial disorders. According to the literature review, the prevalence of PID on thoracic CT scan is one-third of patients. Diffuse interstitial pneumopathy is responsible for a significant morbidity and mortality, is currently under-diagnosed and its treatment is poorly codified. The lung seems to have a central role in the genesis of rheumatoid arthritis. It also appears that some subtypes of anti citrullinated peptide antibodies are preferentially present in the lungs.

The hypothesis behind our project is that one or more subtypes of anti citrullinated peptide antibodies with a preferential tropism for the lung would attack the parenchyma and pulmonary airways.

Currently, there are no data on interstitial pneumopathy in black and Afro-Caribbean subjects with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with rheumatoid arthritis ACR/EULAR 2010
* Patient with a higher age or equal to 18
* Patient receiving social security
* Patient giving his free and informed written consent

Exclusion Criteria:

* Patient with overlap syndrome with another autoimmune disease
* Patients with known severe cardiopulmonary pathology
* Woman who is pregnant and breast feeding
* Patient with language difficulties or understanding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis with diffuse insterstitial lung disease
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Frequency of the positivity of the anti citrullinated peptide antibodies and subtype | three years
  Presence of one or more subtypes of anti citrullinated peptide antibodies in the serum of patients with interstitial pneumopathy associated with rheumatoid arthritis who would be absent

SECONDARY OUTCOMES:
Genetic analysis of the main mutations | three years
  Presence of mutation TERT, RTEL1, PARN et SFTPC

CONTACTS AND LOCATIONS:
Overall Officials: BLETTERY Marie, MD, Principal Investigator — CHU de Martinique
Locations (1):
- CHU Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: Undecided